CLINICAL TRIAL: NCT00127881
Title: Open Label, Dose Escalation, Followed by Open Label,Single Arm Clinical Trial of HuMax-CD4 in Patients With Mycosis Fungoides Type CTCL (Stage IB-IVB) or Sezary Syndrome Who Are Refractory or Intolerant to Targretin® (Bexarotene) and One Other Standard Therapy
Brief Title: Study of Human Monoclonal Antibody to Treat Mycosis Fungoides and Sezary Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: New sponsor, other treatments available
Sponsor: Emergent Product Development Seattle LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hx-CD4-110
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Mycosis Fungoides; Sezary Syndrome
Keywords: Refractory or intolerant to Mycosis Fungoides and sezary syndrome; Cutaneous T-cell Lymphoma; To evaluate the efficacy and safety of zanolimumab in Mycosis Fungoides and sezary syndrome
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — zanolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zanolimumab (Experimental)
  Interventions: Drug: HuMax-CD4 (zanolimumab)

INTERVENTIONS:
Drug: HuMax-CD4 (zanolimumab) — Monoclonal Antibody, 12 weekly infusions.

SUMMARY:
The purpose of this study is to determine the efficacy of the drug, HuMax-CD4, in patients with mycosis fungoides(MF) and sezary syndrome who are intolerant to or do not respond to treatment with Targretin® and one other standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* A biopsy compatible with the diagnosis of MF and sezary syndrome with a CD4 positive phenotype within 6 months of study entry
* Refractory to or intolerant to at least two prior therapies, one being Targretin® (or combinations hereof).
* Signed informed consent

Exclusion Criteria:

* Prior treatment with Total Skin Electron Beam (TSEB) therapy within six months
* Prior treatment with Campath (alemtuzumab)
* Prior treatment with more than three regimens of single agent chemotherapy
* Prior treatment with pentostatin within 6 months
* Treatment within 4 weeks prior to visit 2 with topical Targretin®, skin directed therapies or systemic anticancer therapies, such as, but not limited to: Targretin® , UV-light therapy, local Electron Beam Therapy (EBT), extracorporal photo chemotherapy, methotrexate, bleomycin, cyclophosphamide, combination chemotherapy, oral retinoids, systemic glucocorticosteroids , carmustine, nitrogen mustard, systemic vitamin A or etretinate
* Treatment with topical glucocorticosteroids within 2 weeks prior to visit 2
* Unwillingness or inability to avoid prolonged exposure to the sun or UV light sufficient to produce a mild erythema or thought by the investigator to likely modify the patient's disease
* Concurrent or previous malignancies within the past five years except adequately treated in situ carcinoma of the uterine cervix or basal or squamous cell skin carcinoma
* Significant concurrent, uncontrolled, or active medical condition including, but not limited to renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, cerebral or psychiatric disease
* Known or suspected positive serology for HIV
* Known or suspected positive serology for hepatitis B or C
* Patients who are currently participating in any other trials or having received treatment with any experimental agent within 4 weeks prior to visit 1 (screening)
* Prior treatment with anti-CD4 monoclonal antibodies
* Breast feeding women or women with a positive pregnancy test at Visit 1
* Women of childbearing potential not willing to use either hormonal birth control, an intrauterine device or double-barrier method for the entire study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-07; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
PGA Score | Duration of Study

CONTACTS AND LOCATIONS:
Locations (35):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Tulane University Health Science Center, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - New York Medical Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Middle Tennessee Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- France (4):
  - Hopital de I'Hotel-Dieu, Lyon
  - Consultation Dermatologie Niveau moins 1 Hopital Archet 2, Nice
  - Hopital Saint-Louis Service de Dermatologie, Paris
  - Centre Hospitalier Lyon Sud Bat. 1F 1er etage service Hematologie, Pierre-Bénite
- Germany (5):
  - Skin Cancer Center Charite Mitte Dermatologie Fran Ramona Kursawa, Berlin
  - University of Essen - Universitatsklinikum Essen z. Hd. Frau Desire Zieling, Essen
  - University of kiel, Klinik Fur Dermotologie, Christian-Albrechts-Universitat Zu, Kiel
  - Klinikum Minden / Hautklinik Minden, Minden
  - University of Wurzburg - Universitatsklinikum Wurzburg dermato-onkologische studien, Würzburg
- Italy (5):
  - Instituto di Ematologia e Oncologia Medica "L. & A. Seragnoli", Bologna
  - Day Hospital Oncologico-Presidio Ospedaliero Firenze Centro Ospedale Santa Maria Nuova Azienda Sanitaria di Firenze, University of Florence, Florence
  - University of Milan-Fondazione IRCCS di Natura Pubblica Ospedale Maggiore Policlinico Mangiagalli e Regina Elena di Milano via Francesco Sforza, Milan
  - Instituto Dermopatico dell'Immacolata IRCCS via Monti di Creta, Roma
  - University of Turin SCDU Dermosifilopatia 2 A.S.O. Molinette S.Giovanni Battista, Turin
- Spain (2):
  - Hospital Universitario de la Princesa, Madrid
  - Maternidad Planta Baja, Hospital 12 de Octubre, Madrid